CLINICAL TRIAL: NCT06221800
Title: A Pilot Study to Assess the Diversity of Gut Microbiome in Metastatic Non-Small Cell Lung Cancer (NSCLC) in Correlation to Treatment Effects and Adverse Effects
Brief Title: Assess Diversity of Gut Microbiome in Met NSCLC in Correlation to Tx & Adverse Effects
Status: Recruiting | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Misako Nagasaka, Associate Clinical Professor, University of California, Irvine
Other Study IDs: 3887; UCI 22-86 (Other: UCI CFCCC)
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Microbiota

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Treatment with PD1/L1 monotherapy
  Interventions: Diagnostic Test: Microbiome
- Treatment with PD1/L1 + chemotherapy
  Interventions: Diagnostic Test: Microbiome
- Treatment with Tyrosine Kinase Inhibitor
  Interventions: Diagnostic Test: Microbiome

INTERVENTIONS:
Diagnostic Test: Microbiome — Stool and saliva samples will be collected

SUMMARY:
This is a pilot study collecting data on the diversity and composition of gut microbiomes in subjects with advanced/metastatic Non-Small Cell Lung Cancer (NSCLC) while receiving treatment for NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* 1. Advanced/Metastatic non-small cell lung cancer NSCLC patients.
* 2. The patient himself/herself must be 18 years of age on day of signing informed consent.
* 3. The subject has signed the informed consent form.
* 4. The patient must be eligible to receive FDA approved and non-approved PD1 inhibitors (i.e. pembrolizumab, nivolumab) or PDL1 inhibitor (i.e. atezolizumab, durvalumab) either single agent or as combination therapy with chemotherapy, or be eligible to receive FDA approved and non-approved tyrosine kinase inhibitors.
* 5. The subject will be registered upon submission of the samples. When submitted on separate dates, the submission occurring later will be considered the date of registration

Exclusion Criteria:

* 1. Those subjects who are determined clinically unstable of the participation of this study as determined by the PI or treating physician will be excluded and asked to focus on their treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with advanced/metastatic non-small cell lung cancer (NSCLC)
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Gut microbiomes in advanced/metastatic NSCLC patients | Up to 2 years
  To summarize the diversity and composition of gut microbiomes at baseline or prior to initiation of therapy

SECONDARY OUTCOMES:
Change in microbiome diversity and composition from baseline (prior to start of therapy) to first post-treatment evaluation scan. | Up to 2 years
  Relative difference (and if necessary, relative ratio) between baseline and the first post-evaluation scan
Clinical Response Rate (RR) | Up to 2 years
  Defined according to RECIST v1.1 criteria
Progression-Free Survival (PFS) | Up to 2 years
  Duration from the start date of treatment to the date of progression or death from any cause, whichever occurs first.
Overall survival (OS) | Up to 2 years
  Duration from the start date of treatment to the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Misako Nagasaka, MD,PhD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center University of California, Irvine, Orange, California, United States